CLINICAL TRIAL: NCT06440174
Title: Understanding the Variation of Modern Endoscopic Ultrasound Use in Patients with Oesophageal Cancer (VALUE): a Multi-methods Study
Brief Title: Understanding the Variation of Modern Endoscopic Ultrasound Use in Patients with Oesophageal Cancer (VALUE)
Acronym: VALUE
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: CAN1794
Record Dates: First submitted 2024-05-08; First posted 2024-06-03 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Oesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: endoscopic ultrasound — EUS is an invasive procedure combining upper gastrointestinal endoscopy with ultrasonography. An ultrasound probe located at the end of the endoscope allows direct visualisation of the oesophageal wall layers and adjacent tissues providing local assessment of the depth of tumour invasion and lymph nodes. This assessment informs local tumour (T-) and node (N-) staging which are important prognostic indicators of survival. Patients undergoing EUS require sedation and there are risks of complication. EUS is a specialist investigation requiring many years of dedicated training to perform competently.

SUMMARY:
This is an observational trial that will look at patients undergoing endoscopic ultrasound (EUS) in patients with oesophageal cancer and to determine the proportion of cases in which EUS changes disease management in these patients.

DETAILED DESCRIPTION:
Over 9,000 patients are diagnosed with oesophageal cancer in the United Kingdom (UK) annually. The prognosis of these patients is poor, with an overall 5-year survival rate of 15%.

Most patients (60%) present with advanced disease and palliation is the only treatment option. Accordingly, oesophageal cancer has considerable unmet research need.

The VALUE trial is a prospective observational study investigating EUS in the modern era of oesophageal cancer staging. A quantitative study component will examine how often and why EUS changes treatment decisions after initial staging with CT and PET-CT. A qualitative study component will explore both clinician and patient attitudes and opinions towards the utility of EUS in the staging pathway.

EUS is an invasive procedure combining upper gastrointestinal endoscopy with ultrasonography. An ultrasound probe located at the end of the endoscope allows direct visualisation of the oesophageal wall layers and adjacent tissues providing local assessment of the depth of tumour invasion and lymph nodes. This assessment informs local tumour (T-) and node (N-) staging which are important prognostic indicators of survival. Patients undergoing EUS require sedation and there are risks of complication. EUS is a specialist investigation requiring many years of dedicated training to perform competently.

VALUE aims to recruit patients with oesophageal cancer who are deemed to have potentially curable disease and who are fit for, and wish to have, radical treatment, and who receive EUS as part of their standard of care staging pathway. Patients with a range of disease status (T1-T4; N0-N3) will be considered for recruitment to allow diverse consideration of the reasons whether EUS impacts treatment decisions in current clinical practice. VALUE will also recruit clinicians who regularly care for oesophageal cancer patients in a multi-disciplinary setting to gather their opinions regarding the use of EUS in this patient population.

A systematic review, updating a prior review, found that current evidence concerning the impact of EUS on the management and outcome of oesophageal cancer patients in modern staging with PET-CT was of limited quality. In total, 18 studies with 11,836 patients were included. Overall, 2,805 patients (23.7%) underwent EUS compared to 9,031 (76.3%) without. However, only 19.7% of all patients also had PET-CT for staging. Reported change of management by EUS varied widely from 0% to 56%.

EUS use in oesophageal cancer patients across the NHS is also reported to vary widely. Considerable variation in EUS practice was found in a survey of oesophageal cancer multi-disciplinary team (MDT) leads across the UK. Eighty-seven of 97 UK NHS trusts responded. 29% recommended EUS for all potentially curable patients whereas 46% requested EUS after PET-CT on a case-by-case basis. 20% reported both a lack of utility and concerns about treatment delay. Overall, 63% and 43% routinely use EUS for radiotherapy and surgical planning, respectively. Further, data from the National Oesophago-Gastric Cancer Audit (NOGCA) all describe the reported decline in EUS use from 62% of all patients in 2013, to 39% in 2019, and 18.6% to 2021. In 2020/21, EUS was used in 23.6% of patients who had a curative treatment plan.

The Cancer of Oesophagus or Gastricus-New Assessment of Technology of Endosonography (COGNATE) trial randomised patients between EUS with CT, and CT alone. EUS led to improved quality-adjusted survival. However, since COGNATE, oesophageal cancer staging has been transformed by PET-CT, a cross-sectional nuclear imaging test usually performed prior to EUS. PET-CT has greater sensitivity for distant metastases than CT, and therefore identifies more patients unsuitable for radical treatment, meaning that local staging with EUS becomes less critical in these patients.

This conclusion is supported by data from a large retrospective cohort study by Findlay et al which included 953 patients, of which 798 had EUS, and 918 had PET-CT. The authors found that patient management was changed by EUS in 11% of cases, but when probability thresholds were calculated, the utility of EUS in the majority of patients (71.8% staged T2-T4a) was minimal (0.4%), concluding that the risk of EUS exceeded its benefit. However, these data have not been validated outside of this single-centre study but does question the value of EUS in the modern staging pathway.

In summary, the use of PET-CT for oesophageal cancer staging is increasing, and use of EUS declining, which supports the modern tendency of clinicians to favour non-invasive cross-sectional imaging. However, evidence supporting the basis for this recent change in practice is limited.

There will also be a qualitative part of the trial where a qualitative researcher will interview 30 patients who consent to this in the patient information sheet and 30 clinicians who can carry out EUS, and ask both for their opinions and thoughts on the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 16 or above with first diagnosis of biopsy-confirmed oesophageal cancer.
2. Referred for EUS examination as part of standard of care investigations.
3. Tumour location in the oesophagus, or gastro-oesophageal junction (Siewert types I-III)
4. MDT decision that patient is potentially curable with radical treatment (e.g., endoscopic treatment, surgery +/- neoadjuvant therapy, or definitive chemoradiotherapy)
5. Prior staging with CT and PET-CT
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. Clinical staging of T1-T4, N0-N3, M0 disease
8. Adenocarcinoma or squamous cell carcinoma (SCC) histopathological cell type

   Exclusion Criteria:
9. Recurrent or residual disease
10. Distant metastatic disease detected before EUS.
11. Previous oesophagectomy or oesophageal radiotherapy
12. Unable to undergo EUS examination.
13. Concurrent malignancy e.g., second primary tumour
14. Other histopathological cell type

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited through MDTs at participating secondary care centres in the UK. Those deemed suitable will be approached by their care team to take part.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients who change treatment management | this decision will be made at baseline.
  to determine if using EUS after CT-PET changes management.

SECONDARY OUTCOMES:
Number of clinicians and patients who will share their opinions on EUS by a one to one interview with a qualitative researcher. | This will take place up to 6 weeks following the EUS at one to one interviews.
  The voluntary one to one interview which patients will consent to on the informed consent form, will be used to identify factors that patients consider when deciding whether EUS should be used. This will take place on Microsoft Teams, hosted by the SCTU qualitative researcher. The interview will be recorded and accurately transcribed and once this has taken place, the interview will be deleted. The anonymised transcript can be stored for up to 10 years with the University of Southampton research data management policy.
Number of patients who changed their treatment management following EUS. | this decision will be made at baseline.
  to determine the reasons why EUS changed management.
Number of patients who decided on their treatment. | this decision will be made at baseline.
  to determine the time from diagnosis to treatment decision before and after EUS.

CONTACTS AND LOCATIONS:
Overall Officials: Kieran Foley, Principal Investigator — Chief Investigator, based at Velindre University NHS Trust
Locations (8):
- United Kingdom (8):
  - Royal Bournemouth Hospital, Bournemouth
  - Cambridge University NHS Foundation Trust, Cambridge
  - Velindre University NHS Trust, Cardiff
  - Glasgow Royal Infirmary, Glasgow
  - Castle Hill Hospital, Hull
  - Imperial College Healthcare NHS Trust, London
  - University Hospital Southampton, Southampton
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foley KG, Boxall C, Franklin J, Cook A, Underwood T, Griffiths G, Cozens K, Bradbury K, Fay M, Chuter D, Longman KA, Lindfield B, Hurt C. Understanding the variation of modern endoscopic ultrasound use in patients with oesophageal cancer (VALUE): protocol for a multi-methods study. BJR Open. 2025 May 21;7(1):tzaf012. doi: 10.1093/bjro/tzaf012. eCollection 2025 Jan. PMID 40486070